CLINICAL TRIAL: NCT00072943
Title: A Phase II, Double-Blind, Placebo-Controlled Study to Determine the Safety and Efficacy of a Humanized Anti-Interferon-γ Monoclonal Antibody (HuZAF) Administered to Patients With Moderate to Severe Crohn's Disease
Brief Title: A Humanized Anti-Interferon-γ Monoclonal Antibody (HuZAF) for Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Facet Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 707
Record Dates: First submitted 2003-11-12; First posted 2003-11-17 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Crohn's Disease; Colitis; Intestinal Disease; Gastrointestinal Disease; Digestive System Disease
Keywords: Crohn's Disease; Colitis; Monoclonal antibody therapy; anti-interferon gamma
MeSH Terms: conditions — Crohn Disease; Colitis; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases

INTERVENTIONS:
Drug: anti-Interferon-gamma monoclonal antibody

SUMMARY:
The purpose of the HARMONY study is to assess the safety and efficacy of an investigational drug called HuZAF, in patients with moderate to severe Crohn's disease (CD). HuZAF is a humanized anti-Interferon-gamma (anti-IFN-γ) monoclonal antibody, which binds and blocks IFN-γ, a protein in the immune system that is involved in inflammation. Antibodies are proteins normally produced by our immune system to help fight off foreign substances. Scientists have been able to make therapeutic humanized monoclonal antibodies, similar to the antibodies in our bodies, to target diseases.

DETAILED DESCRIPTION:
Participants will be randomized, assigned by chance, to one of five treatment groups consisting of: four groups differing in the amount of study drug given and one placebo group. The initial dose of study drug will be given intravenously, injected into a vein in the arm. Four weeks later, three subsequent doses of study drug will be given subcutaneously, through the skin, every four weeks for three doses. Patients will be followed for approximately six months after receiving their final dose.

ELIGIBILITY:
* Patients 18-70 years old
* Patients with moderate to severe Crohn's disease
* Patients who have had Crohn's disease for at least 6 months
* Patients who have previously been treated for Crohn's disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175
Dates: Start 2002-03; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (15):
  - Advanced Clinical Research Institute, Anaheim, California
  - Doctor's Office, Orange, California
  - Gainesville VA Medical Center, Gainesville, Florida
  - Waterside Clinical Research Services, Inc., West Palm Beach, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Doctor's Office, Chicago, Illinois
  - University of Kentucky Medical Center, Division of Digestive Disease & Nutrition, Lexington, Kentucky
  - Massachusetts General Hospital, Gastrointestinal Unit, Boston, Massachusetts
  - Gastroenterology Specialities P.C., Lincoln, Nebraska
  - Carolina Digestion Health Associates, Charlottesville, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University Pittsburgh Medical Center, Division of Gastroenterology, Hepatology and Nutrition, Inflammatory Bowel Disease Center, Pittsburgh, Pennsylvania
  - Houston Medical Research Associates, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Canada (4):
  - Vancouver General Hospital, Dept. of Medicine, Vancouver, British Columbia
  - Health Science Centre, Winnipeg, Manitoba
  - Queen Elizabeth II Health Science Center, McKenzie Building, Pathology, Halifax, Nova Scotia
  - London Health Science Center, University Campus, London, Ontario

REFERENCES:
- See also: Crohn's and Colitis Foundation of America — http://www.ccfa.org
- See also: Harmony Study — http://www.harmonystudy.com